CLINICAL TRIAL: NCT03715959
Title: Phi29 Motor Nanopore for Single Molecule Sensing: Breast Nipple Aspirate Fluid
Brief Title: Nipple Aspirate Fluid in Detecting Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, William Carson, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-16288; NCI-2018-01437 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Estrogen Receptor Negative; Healthy Subject; HER2 Positive Breast Carcinoma; HER2/Neu Negative; Luminal A Breast Carcinoma; Luminal B Breast Carcinoma; Progesterone Receptor Negative; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (nipple aspiration fluid) (Experimental): Participants and healthy volunteers undergo collection of nipple aspirate fluid from both breasts.
  Interventions: Procedure: Aspiration of Breast; Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Aspiration of Breast — Undergo NAF
Procedure: Biospecimen Collection — Undergo NAF

SUMMARY:
This trial studies nipple aspirate fluid in detecting breast cancer. Nipple aspirate fluid may better detect breast cancer earlier than current methods used for screening such as mammograms and breast examinations.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain nipple aspirate fluid (NAF) samples from non-lactating women subjects at least 40-years-old.

II. To analyze the samples using a novel protein nanopore-based detection platform to evaluate the efficacy of the platform for breast cancer diagnosis through detection of biomarkers.

OUTLINE:

Participants and healthy volunteers undergo collection of nipple aspirate fluid from both breasts.

After completion of study, participants are followed up at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* BREAST CANCER: Must be > 1 year from pregnancy, lactation.
* BREAST CANCER: Must be currently diagnosed with known breast cancer in breast.
* BREAST CANCER: Must not be currently diagnosed with cancers other than breast cancer.
* BREAST CANCER: Must not have been gone through surgery, radiotherapy or chemotherapy within 30 days of enrollment.
* HEALTHY SUBJECTS: No history of breast cancer and must not be currently diagnosed with any other cancer.
* HEALTHY SUBJECTS: Must be > 1 year from pregnancy, lactation.
* HEALTHY SUBJECTS: Must be willing to have a clinical breast exam and/or mammogram performed or reviewed by an Ohio State University (OSU) radiologist at the James Cancer Hospital within the past 90 days prior to their NAF procedure. The clinical breast exam result and/or mammograms must be read as not suspicious for breast cancer.
* HEALTHY SUBJECTS: Must be willing to keep the clinic informed of their breast health status for 1 year.

Exclusion Criteria:

* Subjects who are currently pregnant, lactating, or within a year of pregnancy/lactation. Pregnancy testing will not be required of any patients over 60 years of age, or any patient who has undergone bilateral oophorectomy.
* Subjects who currently are diagnosed with cancers other than breast cancer.
* Subjects who cannot give an informed consent.
* Male gender of any age.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Biomarkers expression levels | Up to 1 year
  Nipple aspiration fluid samples will be compared between breast cancer participants and healthy participants. will perform the logistic regression model for each biomarker that shows any difference between the breast cancer patients and healthy individuals. Then we will include multiple biomarkers in one model while controlling for confounders.

CONTACTS AND LOCATIONS:
Overall Officials: William Carson, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu